CLINICAL TRIAL: NCT02552810
Title: Effect of Plasma of Argon Cleaning on Implant Abutments in Patients With a History of Periodontal Disease and Thin Biotype: Five Years Post-loading Results of a Randomized Controlled Trial
Brief Title: Plasma of Argon Cleaning on Implant Abutments: 5-year Results of a Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Luigi Canullo, Clinical researcher, study adviser, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UValencia_001_Plasma
Record Dates: First submitted 2015-09-14; First posted 2015-09-17 (Estimated); Results first posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-05

CONDITIONS: Endosseous Dental Implant Failure; Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Plasma of Argon (Active Comparator): Abutment cleaning by plasma of Argon protocol .
  Interventions: Device: Plasma of Argon
- Steam clean (Active Comparator): Abutment cleaning by steam clean device.
  Interventions: Device: Steam clean

INTERVENTIONS:
Device: Steam clean — Control group: dental implant abutments underwent cleaning by steam (VAP 1, Zhermark, Cologne, Germany), performed for 5 seconds at 4 megapascal (MPa).
  Arms: Steam clean
Device: Plasma of Argon — Test group: dental implant underwent argon plasma treatment in a plasma reactor (Diener Electronic, Jettingen, Germany). The treatment conditions were 75 W of power and 1 bar of pressure for 12 minutes.
  Arms: Plasma of Argon

SUMMARY:
Contamination of implant abutments could potentially influence the peri-implant tissue inflammatory response. The aim of the present study was to assess the radiographic bone changes around customized, platform switched, abutments placed according to the "one-abutment-one-time" protocol, with and without plasma of argon cleaning treatment.

DETAILED DESCRIPTION:
After technical procedures, presence of contaminants (mostly Titanium wear micro-particles, Carbon and Aluminum traces due to lubricant used during customization) on the whole abutment surface, the internal connection and the screw can be found, even after the usually cleaning steps (steaming).

Such debris, present at titanium/connective-bone tissues interface (gingival portion of the abutment), could directly or indirectly deleteriously influence the inflammatory response on the peri-implant tissues.

Plasma of Argon cleaning treatment was demonstrated to have a double effect on titanium abutments: removal of pollutions following customization and increase of cell adhesion. Additionally, Plasma of Argon demonstrated very potent anti-biofilm activity. This prospective, match paired, triple-blinded randomized controlled trial was aimed to test if plasma treatment of customized abutments can affect radiographic peri-implant marginal bone level changes after 5 years of prosthetic loading.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older, previously treated for periodontal disease according to a comprehensive treatment strategy,25 requiring a single implant-supported restoration in the anterior maxilla or premolar region with the presence of mesial and distal tooth.
* Bone crest allowing the insertion of a 4 mm platform implant without further bone augmentation procedures and with thin (≤ 1 mm) gingival biotype, measured by previously reported protocol.

Exclusion Criteria:

* no relevant medical conditions;
* non-smoker or smoking ≤ 10 cigarettes/day;
* plaque Index and bleeding on probing ≤ 25 %;
* impossibility of follow-up for 5 years after prosthetic loading;
* pregnant and lactating patients;
* patients with a history of bisphosphonate therapy;
* presence of sites with acute infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Canullo, Principal Investigator — University of Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Canullo L, Penarrocha D, Clementini M, Iannello G, Micarelli C. Impact of plasma of argon cleaning treatment on implant abutments in patients with a history of periodontal disease and thin biotype: radiographic results at 24-month follow-up of a RCT. Clin Oral Implants Res. 2015;26(1):8-14. doi: 10.1111/clr.12290. Epub 2013 Nov 6. PMID 24191873

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients who met the inclusion criteria were asked to participate and were enrolled in consecutive order between January and September 2010 at the Department of Oral Surgery, University of Valencia.
Groups:
- Plasma of Argon: Abutment cleaning by plasma of Argon protocol .
  Dental implant placement: Using a surgical stent, patients received one implant in the anterior or premolar region of the maxilla.
  Second stage surgery: After 3 months of healing, a minimally invasive flap for the second surgery procedure was performed.
  Abutment connection: Abutments were randomly allocated to control (subjected only to the usually adopted steam cleaning) and test groups (subjected to plasma of argon cleaning).
  Plasma of Argon: Test group abutments underwent argon plasma treatment in a plasma reactor (Diener Electronic, Jettingen, Germany). The treatment conditions were 75 W of power and 1 bar of pressure for 12 minutes.
- Steam Clean: Cleaning protocol by steaming.
  Dental implant placement: Using a surgical stent, patients received one implant in the anterior or premolar region of the maxilla.
  Second stage surgery: After 3 months of healing, a minimally invasive flap for the second surgery procedure was performed.
  Abutment connection: Abutments were randomly allocated to control (subjected only to the usually adopted steam cleaning) and test groups (subjected to plasma of argon cleaning).
  Steam cleaning: Control group abutments underwent cleaning by steam (VAP 1, Zhermark, Cologne, Germany), performed for 5 seconds at 4 MPa.
Period: Overall Study
Arm/Group | Plasma of Argon | Steam Clean
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Test Group: Test group abutments, after milled, polished and cleaned for 30s in the same laboratory, underwent argon plasma treatment (75 W of power and -10 MPa of pressure for 12 minutes at room temperature) in a plasma reactor8 located in the same clinic but in a different room. All the abutments were then handed to the clinician in a sterile envelope, without the possibility to evaluate the treatment undergone.
- Control Group: Control group were cleaned by steam for 30s 7 by the dental technician in the laboratory located in the same clinic, but in a different room, immediately before delivering to the clinician. Then all the abutments were then handed to the clinician in a sterile envelope, without the possibility to evaluate the treatment undergone.
- Total: Total of all reporting groups
Arm/Group | Test Group | Control Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Full Range); unit: years] | 56.3 [31 to 77] | 60.1 [37 to 79] | 58.4 [31 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  Spain | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Success Rate of the Implants and Prostheses (Participants).
Description: An implant was considered a failure if it presented any mobility, assessed by tapping or rocking the implant head with the metallic handles of two instruments, and/or any signs of radiolucency, progressive marginal bone loss or infection, and any mechanical complications (e.g. implant fracture) rendering the implant unusable, though still mechanically stable in the bone. This was evaluated on an intraoral radiograph taken with a paralleling technique strictly perpendicular to the implant-bone interface. The implant stability was assessed at initial loading and following 3 years of application, with the prostheses removed.
  A prosthesis was considered a failure if it needed to be replaced by an alternative prosthesis.
Time Frame: During all the follow-up (5 years)
Measure: Number; unit: percentage of participants
Arm/Group | Plasma of Argon | Steam Clean
Number analyzed (Participants) | 15 | 15
percentage of participants | 100 | 100
Statistical Analysis 1: Comparison: Plasma of Argon vs Steam Clean; Test type: Non-Inferiority or Equivalence — Sample size calculation, 30 (effect size: 0.5, alpha error: 0.05, power: 0.80); p < 0.05, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Any Biological or Technical Complications.
Description: Complications: any biological (pain, swelling, suppuration, etc) and/or mechanical complications (fracture of the framework and/or the veneering material, screw loosening, etc) were considered.
Time Frame: During all the follow-up (5 years)
Measure: Number; unit: participants
Arm/Group | Plasma of Argon | Steam Clean
Number analyzed (Participants) | 15 | 15
participants | 0 | 0

3. Secondary Outcome: Peri-implant Marginal Bone Level Changes (Express in mm).
Description: At the time of loading with the provisional crown (T0), periapical standardized digital or analogical radiographs were taken in order to control the perfect adaptation of the abutment on the implant and control peri-implant bone level. The customized film holder was made using an hard silicone on the bite of film holders (Rinn XCP; Dentsply Rinn, Elgin, IL, USA) and the parallel technique was used. Radiographs were also taken at 12 (T1), 24 (T2), 48 (T4), and 60 months (T5) after the final restoration delivery, to evaluate marginal bone level changes.
Time Frame: At 5 years.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Plasma of Argon | Steam Clean
Number analyzed (Participants) | 15 | 15
mm | 0.21 (0.21) | 0.65 (0.36)

4. Secondary Outcome: Esthetic Parameters Measured as the Changes in Mesial and Distal Papilla Height (PH) and Buccal Peri-implant Mucosa Changes at the Zenith (REC), Expressed in mm.
Description: A customized millimeter tubular support (stent) was placed temporarily around each dental implant. For each site, mesial and distal soft tissue dimensions (papilla height, PH), and buccal peri-implant mucosa dimension at the zenith (REC) were measured, and reported in millimeters. Two measurements were recorded. The first at definitive crown delivery (baseline), and the second at the 5 years follow-up examination. Changes in PH and REC were reported in millimeters as the difference between values recorded at the 5-year follow-up and the baseline.
  The full procedure was published in:
  Canullo L, Iurlaro G, Iannello G. Double-blind randomized controlled trial study on post-extraction immediately restored implants using the switching platform concept: soft tissue response. Preliminary report. Clinical Oral Implants Research [Internet]. 2009 Apr;20(4):414-20.
Time Frame: At 5 years.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Plasma of Argon | Steam Clean
Number analyzed (Participants) | 15 | 15
mm
  PH | 0.48 (0.40) | 0.39 (0.31)
  REC | 0.58 (0.66) | 0.22 (0.35)

5. Secondary Outcome: Percentage of Patients With Plaque Index
Description: Modified Plaque Index (mPI) was evaluated as the amount of plaque at the cervical part of the implant-supported crown, scored by running a probe along the implant-supported crown surface. Measured as Yes or Not.
Time Frame: At 5 years.
Measure: Number; unit: percentage of participants
Arm/Group | Plasma of Argon | Steam Clean
Number analyzed (Participants) | 15 | 15
percentage of participants | 13.3 | 13.3

6. Secondary Outcome: Percentage of Patients With Bleeding on Probing
Description: Presence of bleeding within 10 seconds after probing. Measured as Yes or Not.
Time Frame: At 5 years.
Measure: Number; unit: percentage of participants
Arm/Group | Plasma of Argon | Steam Clean
Number analyzed (Participants) | 15 | 15
percentage of participants | 6.6 | 20

ADVERSE EVENTS:
Time Frame: Five years (during all the follow-up).
Description: Radiographs at 6-, 12-, 24-, 48-, and 60 months after function. Periodontal parameters every six months. Aesthetic at baseline and 5 years later.
Arm/Group | Plasma of Argon | Steam Clean
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No